CLINICAL TRIAL: NCT06695052
Title: "Axillary Nodal Evaluation in Breast Cancer by Multimodal US"
Brief Title: Axillary LNs Evalution in Breast Cancer by Multimodal Us
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Heba Abo Elmakarem Ahmed, doctor, Assiut University
Other Study IDs: Axillary LNs in BC by multi US
Record Dates: First submitted 2024-11-05; First posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Lymph Node Metastasis
Keywords: breast cancer; Lymph Node Metastasis; multimodal ultrasound
MeSH Terms: conditions — Breast Neoplasms; Lymphatic Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: multi modal Us — Greyscale US: grey scale ultrasound Color Doppler US: Color Doppler ultrasound Elastography US: Elastography ultrasound

SUMMARY:
The present study is designed to evaluate the role of simultaneous multi-modal sonographic tools-Ultrasound (US), Color Doppler Ultrasound (CDU), and Ultrasound Elastography (UE)-in determining the nature (benign or malignant) of axillary lymph nodes (ALNs) in patients with primary breast cancer. It aims to compare the diagnostic indices of each modality individually against their combined performance. Specifically, the study will assess whether adding UE to conventional gray-scale US and CDU improves diagnostic accuracy.

DETAILED DESCRIPTION:
Breast cancer (BrCa) is the most common malignant tumor affecting women globally, with its incidence and cancer-related mortality rates continuing to rise. Accurate evaluation of the presence, extent, and status of ALNs is critical for prognosis, disease staging, and treatment planning in patients with breast cancer.

Historically, axillary lymph node dissection (ALND), followed by histopathological evaluation, was the standard method for staging breast cancer. However, ALND is associated with short- and long-term complications such as lymphedema, nerve injury, seroma formation, and infection. To reduce these risks, sentinel lymph node biopsy (SLNB) has largely replaced ALND. While SLNB is less invasive and has fewer complications, it is still associated with a risk of false-negative results. According to the American Society of Oncology Guidelines, if SLNB results are negative, no further ALND is performed, as it does not confer a survival benefit. Patients with positive SLNB results, however, undergo a "completion" ALND.

Role of Ultrasound and Color Doppler Ultrasound:

Gray-scale ultrasound (US) is a non-invasive imaging modality widely used for the preoperative evaluation of ALNs in breast cancer patients. It provides valuable morphological information and facilitates obtaining tissue samples. However, its diagnostic accuracy is operator-dependent and limited to structural features of the lymph nodes. Adding Color Doppler Ultrasound (CDU) enhances this evaluation by providing functional insights, such as assessing vascular patterns and calculating the resistive index (RI) of ALNs. Despite their potential, US and CDU exhibit highly variable sensitivity and specificity across studies, which limits their standalone diagnostic utility.

Role of Ultrasound Elastography (UE):

Real-time strain ultrasound elastography (UE) is an advanced imaging technique that measures tissue stiffness, a property often associated with malignancy. Unlike US and CDU, UE can quantify stiffness, providing additional diagnostic insights. Elastography utilizes rhythmic manual compression to produce color-coded elastograms, which display differences in tissue stiffness. These elastograms are generated alongside conventional gray-scale US to ensure precise imaging of the same lymph node. Although UE has been explored for ALN assessment, existing studies report inconsistent results.

Recent meta-analyses suggest that UE offers valuable supplementary information for preoperative ALN evaluation and may influence surgical decision-making.

Other Imaging Modalities:

Alternative imaging techniques, including mammography, magnetic resonance imaging (MRI), multi-detector computed tomography (CT), and positron-emission tomography (PET-CT), have also been employed for ALN assessment. However, their widespread application is limited by moderate sensitivity, low specificity, high costs, radiation exposure, and the need for specialized imaging protocols for ALNs.

Multimodal Imaging:

Multimodal imaging, which combines two or more imaging techniques, provides a more comprehensive diagnostic approach than individual modalities alone. This study investigates the combined use of gray-scale US, CDU, and UE to improve diagnostic accuracy for ALN assessment in breast cancer patients.

This version addresses the study's purpose, methodology, and the role of each modality in greater detail

ELIGIBILITY:
Inclusion Criteria:

- Patients with primary breast cancer (BrCa) and axillary lymph nodes (ALNs) referred to the Department of Diagnostic Radiology for pre-operative assessment of presence, extent and nature of ALNs.

Exclusion Criteria:

* Patients with secondary or recurrent Breast Ca
* Patients exposed to loco-regional radio- or chemotherapy
* Patients with previous axilla surgery
* ± Patients with confirmed metastatic tumor to bone, liver and/or lungs
* Patients who deny or refuse to participate in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Female patients with primary breast cancer and metastatic axillary LNs
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-11-20 (Estimated); Primary Completion 2026-11-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Evaluation of axillary LNs in Breast Cancer by Grey Scale Ultrasound | Baseline
  Evaluate axillary lymph nodes (LNs) in breast cancer patients using grey scale ultrasound to assess specific characteristics such as size, shape, and cortical thickening. Results will be compared to Fine Needle Aspiration Cytology (FNAC) or histopathology findings.
Evaluation of axillary LNs in Breast Cancer by Color Doppler Ultrasound | Baseline
  Evaluate axillary lymph nodes (LNs) in breast cancer patients using color Doppler ultrasound to assess vascularity patterns. Results will be compared to FNAC or histopathology findings.
Evaluation of axillary LNs in Breast Cancer by Elastography Ultrasound | Baseline
  Evaluate axillary lymph nodes (LNs) in breast cancer patients using elastography ultrasound to measure stiffness and elasticity. Results will be compared to FNAC or histopathology findings.
Comparison of Multimodal Ultrasound Findings with Histopathology Results | Baseline
  Compare the findings from grey scale ultrasound, color Doppler ultrasound, and elastography ultrasound with histopathology results to assess diagnostic accuracy for evaluating axillary lymph nodes in breast cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Abul Hassan H Mohammed, AP.radiology, Study Director — Assiut University; Sara M Ahmed, AP.radiology, Study Director — Assiut University

REFERENCES:
- [Background] Tsai WC, Lin CK, Wei HK, Yu BL, Hung CF, Cheng SH, Chen CM. Sonographic elastography improves the sensitivity and specificity of axilla sampling in breast cancer: a prospective study. Ultrasound Med Biol. 2013 Jun;39(6):941-9. doi: 10.1016/j.ultrasmedbio.2012.12.013. Epub 2013 Mar 7. PMID 23465139
- [Background] DeSantis CE, Ma J, Gaudet MM, Newman LA, Miller KD, Goding Sauer A, Jemal A, Siegel RL. Breast cancer statistics, 2019. CA Cancer J Clin. 2019 Nov;69(6):438-451. doi: 10.3322/caac.21583. Epub 2019 Oct 2. PMID 31577379